CLINICAL TRIAL: NCT05802485
Title: PANCREATIC CANCER: DYNAMIC ASSESSMENT AT ALL STAGES OF TREATMENT: PANDORE-PANC-IPC 2021-082
Brief Title: PANCREATIC CANCER: DYNAMIC ASSESSMENT AT ALL STAGES OF TREATMENT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PANDORE-PANC-IPC 2021-082
Record Dates: First submitted 2022-11-23; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Pancreatic Cancer Non-resectable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- collection of blood and tumor samples (Other)
  Interventions: Other: collection of blood and tumor samples

INTERVENTIONS:
Other: collection of blood and tumor samples — The study consists of the collection of a 25 ml blood sample:
  * Before the start of treatment
  * Approximately 2 months after the start of induction chemotherapy
  * At the end of induction chemotherapy
  * Prior to local treatment (radiotherapy, surgery)
  * At the time of tumor progression
  At the time of collection of tumor material:
  * During the initial diagnostic biopsy
  * On the operating room in case of surgery
  * During a tumor biopsy in case of recurrence or progression (optional) and a questionnaire evaluating the patient's spontaneous physical activities.

SUMMARY:
The study consists of a 25 ml blood sample collection:

* Before the start of treatment
* Approximately 2 months after the start of induction chemotherapy
* At the end of induction chemotherapy
* Prior to local treatment (radiotherapy, surgery)
* At the time of tumor progression

Collection of tumor material:

* During the initial diagnostic biopsy
* On the operating room in case of surgery
* At tumor biopsy in case of recurrence or progression (optional) As well as the completion of a questionnaire at inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Non-metastatic pancreatic adenocarcinoma that is not immediately resectable (borderline and locally advanced tumors according to the NCCN 2020 classification)
* No previous treatment with surgery or chemotherapy
* Age > 18 years
* General condition WHO 0-2 (patient whose general condition can allow medical treatment or surgery)
* Therapeutic management at the Paoli-Calmettes Institute
* Signature of the informed consent specific to the PANDORE-PANC study
* Patient affiliated to a social security system or benefiting from such a system

Exclusion Criteria:

* Metastatic disease
* Pancreatic tumor of a histological type other than adenocarcinoma
* Other tumor under treatment or for which treatments have been completed for < 1 year
* Pregnant or breastfeeding women
* Person in an emergency situation
* Person of legal age under legal protection (guardianship, curatorship or safeguard of justice) or unable to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Predict response to systemic therapies in patients with non-metastatic pancreatic adenocarcinoma | up to 6 years
  Analysis of the impact of identified biomarkers on overall patient survival and tumour response